CLINICAL TRIAL: NCT01558180
Title: Telephone Care Management to Address Sleep Problems in Young Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: The Ingram Foundation is funding this work. (Unknown)
Responsible Party: Principal Investigator, Jack Stevens, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB11-00719
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Autism Spectrum Disorders; Insomnia
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone Care Management (Experimental): calls from a registered nurse to educate caregivers about behavioral sleep strategies
  Interventions: Behavioral: Telephone Care Management
- Usual Care (Placebo Comparator): It's a placebo comparator because individuals in this group will receive an educational handout on behavioral sleep strategies. This handout approximates standard of care.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telephone Care Management — series of phone calls from registered nurse to discuss behavioral suggestions for pediatric insomnia
  Other Names: TCM
  Arms: Telephone Care Management
Behavioral: Usual Care — educational handouts on pediatric insomnia
  Other Names: UC
  Arms: Usual Care

SUMMARY:
The investigators will conduct a randomized controlled trial comparing a telephone based intervention (TCM) to usual care (UC). TCM will feature a registered nurse providing a series of phone calls to assist caregivers in learning and modifying behavioral strategies that may help young children with autism to sleep better. Objective (activity monitors) and subjective (rating scales) data will be collected by an independent research assistant at the end of the project. The investigators hypothesize that TCM improves sleep duration and decreases sleep problems relative to a usual care control condition (UC).

DETAILED DESCRIPTION:
Please see brief summary.

ELIGIBILITY:
Inclusion Criteria:

1. Insomnia
2. Autism Spectrum Disorder
3. Regular telephone service for caregiver
4. Stable dose of medication

Exclusion Criteria:

1. Signs of obstructive sleep apnea (e.g., turning blue or stop breathing at night, recurrent snoring)
2. Receptive language skills under 18 months

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Children's Sleep Habits Questionnaire | 2 month follow-up

SECONDARY OUTCOMES:
Actigraphy (Activity Monitoring) | 2 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jack Stevens, Ph.D., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States